CLINICAL TRIAL: NCT05039515
Title: A Phase 2 Study to Assess the Efficacy and Safety of 2 Dosage Regimens of Oral Fidrisertib (IPN60130) for the Treatment of Fibrodysplasia Ossificans Progressiva in Male and Female Paediatric and Adult Participants.
Brief Title: A Study to Assess the Effectiveness and Safety of 2 Dosage Regimens of Oral Fidrisertib (IPN60130) for the Treatment of Fibrodysplasia Ossificans Progressiva (FOP).
Acronym: FALKON
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-CA-60130-452; 2020-002858-24 (EudraCT Number); 2024-511469-13-00 (EU CTIS Number)
Record Dates: First submitted 2021-09-02; First posted 2021-09-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Fibrodysplasia Ossificans Progressiva
MeSH Terms: conditions — Myositis Ossificans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IPN60130 high dosage (Experimental): Oral capsule, swallowed whole or sprinkled onto food, once daily
  Interventions: Drug: IPN60130
- IPN60130 low dosage (Experimental): Oral capsule, swallowed whole or sprinkled onto food, once daily
  Interventions: Drug: IPN60130
- Placebo (Placebo Comparator): Oral capsule, swallowed whole or sprinkled onto food, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IPN60130 — Immediate-release capsule containing high dose of the drug substance.
  Other Names: Fidrisertib
  Arms: IPN60130 high dosage
Drug: IPN60130 — Immediate-release capsule containing low dose of the drug substance.
  Other Names: Fidrisertib
  Arms: IPN60130 low dosage
Drug: Placebo — Placebo will be supplied as powder filled hard capsules
  Arms: Placebo

SUMMARY:
Fibrodysplasia Ossificans Progressiva (FOP) is a rare, severely disabling disease characterized by the presence of bone in soft tissue where bone normally does not exist, known as Heterotopic Ossification (HO). It is often associated with painful, recurrent episodes of soft tissue swelling (flare-ups) that lead to abnormal stiffening and immobility (ankyloses) of major joints with cumulative and irreversible loss of movement and disability.

This study will evaluate the efficacy of 2 dosing regimens of IPN60130 in inhibiting new HO volume compared with placebo (a dummy treatment) in adult and paediatric participants with FOP. It will be assessed by a scan (provides internal images of the body) called low dose Whole Body Computed Tomography (WBCT), excluding head.

Adults and participants 5 years of age or older are also eligible for a sub study to evaluate HO lesions assessed by another type of scan, Fluorine-18-labelled natrium fluoride Positron Emission Tomography-Computed Tomography ([18F]NaF PET-CT ).

DETAILED DESCRIPTION:
Note on Primary Completion Date and Results Disclosure:

The Primary Completion Date (PCD) reflects the date when data collection is completed for all primary outcomes, as defined in the Final Rule (42 CFR Part 11). In this study, safety outcomes are designated as primary and collected through the end of study.

Therefore the PCD has been updated to align with this definition. The interim analyses will proceed per the protocol and SAP. Results will be disclosed in line with applicable regulatory timelines.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must be at least 5 years of age, to be confirmed (entry for younger paediatric participants <15 years of age will only be once safety in adult and older paediatric participants ≥15 years of age has been established) at the time of signing the informed participant/parent consent and, for participants who are minors, age-appropriate assent.
* Participants must be at least 15 years of age at the time of signing the informed participant/parent consent for the main study and, for participants who are minors, age-appropriate assent
* Participants must be clinically diagnosed with FOP, with the R206H ACVR1 mutation or other FOP variants associated with progressive HO.
* Participants must have disease progression in the preceding year of the screening visit.
* Participants who have participated in a prior clinical study using another investigational product for the treatment of FOP may be enrolled after a washout of at least 5 half-lives of the other investigational product. Participants with prior treatment such as, but not limited to, imatinib, isotretinoin, garetosmab, or palovarotene may be enrolled 30 days after discontinuation or after washout of at least 5 half-lives, whichever is longer.

  1. Washout period for palovarotene is 30 days
  2. Washout period for garetosmab is 4 months
* Participants must be able to perform pulmonary function tests adequately and reliably.
* Participants must be able to have an adequate echocardiography assessment at screening for evaluation of left ventricular structure and function as defined by the protocol.
* Participants must be accessible for treatment and follow-up and be able to undergo all study procedures. Participants living at distant locations from the investigational site must be able and willing to travel to a site for the initial and all on-site follow-up visits. Participants must be able to undergo low-dose WBCT (excluding head) without sedation.
* Body weight ≥10 kg.
* Abstinent or using two highly effective forms of birth control. Females must also have a negative blood or urine pregnancy test prior to administration of study drug.
* Participants must be capable of giving written, signed, and dated informed participant/parent consent; and for participants who are minors, age-appropriate assent and/or legal guardian consent (performed according to local regulations)

Key Exclusion Criteria:

* Participants with complete heart block and left bundle branch block on screening electrocardiogram.
* Participants with screening echocardiography showing septal or left ventricular free wall thickness >12 mm for adult participants or a z-score >3 compared with population norms for children and adolescent participants or left ventricular ejection fraction (LVEF) <50%.
* Participants with severe mitral or tricuspid regurgitation on echocardiography at screening.
* Participants with significant underlying lung disease requiring supplementary oxygen or forced vital capacity <35% of predicted at screening.
* Participants with uncontrolled cardiovascular, hepatic, pulmonary, gastrointestinal, endocrine, metabolic, ophthalmologic, immunologic, psychiatric, or another significant disease as judged by the investigator.
* Participants with severe hepatic impairment.
* Concomitant medications that are strong inhibitors (including grapefruit juice) or inducers (including St John's Wort) of cytochrome P450 (CYP) 3A4 activity; or kinase inhibitors such as imatinib.
* Prior use in the past year and concomitant use of bisphosphonates for participants in the PET-CT sub study.
* Concurrent participation in another interventional clinical study, or a noninterventional study with radiographic measures or invasive procedures (e.g. collection of blood or tissue samples).
* Amylase or lipase >2× the upper limit of normal (ULN) or with a history of chronic pancreatitis.
* Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5×ULN.
* Participants with hematologic abnormalities:

  * Hgb<10g/dL
  * Platelets<75,000/mm3
  * WBC<2000/mm3

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Annualized change in HO volume as assessed by low-dose WBCT (excluding the head) in treated participants receiving IPN60130 compared with placebo. | From baseline to 12 months
Incidence of Adverse Events / Serious Adverse Events (AEs/SAE) | From baseline until the end of study (63 months)
Change from baseline in clinically significant abnormal values in laboratory parameters (haematology, biochemistry, and urinalysis) | From baseline until the end of study (63 months)
  Percentage of participants with clinically significant change in laboratory parameters (biochemistry, hematology and urinalysis) will be reported. The clinical significance will be graded by the investigator.
Change from baseline in physical examination findings | From baseline until the end of study (63 months)
  Percentage of participants with clinically significant changes in physical examination findings will be reported. The clinical significance will be graded by the investigator.
Change from baseline in clinically significant vital signs | From baseline until the end of study (63 months)
  Percentage of participants with clinically significant changes in Vital Signs will be reported. The clinical significance will be graded by the investigator.
Change from baseline in clinically significant Electrocardiogram (ECG) readings | From baseline until the end of study (63 months)
  Percentage of participants with clinically significant changes in ECG readings will be reported. The clinical significance will be graded by the investigator.

SECONDARY OUTCOMES:
Change in HO volume of new HO lesions as detected by WBCT in participants receiving IPN60130 compared with placebo recipients | From baseline up to 12 months
Change in number of HO lesions by WBCT in participants receiving IPN60130 compared with placebo recipients | From baseline up to 12 months
Flare-up rate and number of flare-up days in participants receiving IPN60130 compared with placebo recipients | From baseline up to 12 months
  The rate and the number of flare-up days, the flare-up being confirmed by the Investigator, will be compared between participants treated with IPN60130 and those treated with Placebo at Month 12
The number of body regions with new HO in participants receiving IPN60130 compared with placebo recipients | From baseline up to 12 months
Change in pain intensity | From baseline up to 12 months
  Assessed in participants ≥13 years old with the Numeric pain rating scale (NRS) and in participants <13 years old with Wong Baker Faces Pain Scale (FPS)
The proportion of participants with any new HO in participants receiving IPN60130 compared with placebo recipients | From baseline up to 12 months
Change from baseline in HO volume as detected by WBCT in participants receiving IPN60130 compared with placebo recipients and with participants receiving the standard of care in the Natural history study (NHS) | From baseline up to 60 months
Change from baseline in Cumulative Analogue Joint Involvement Scale for FOP (CAJIS) by treatment arm compared with placebo recipients and participants receiving the standard of care in the NHS across all available timepoints | From baseline up to 60 months
Change in the FOP Physical Function Questionnaire (FOP-PFQ) by treatment arm compared with placebo recipients and participants receiving the standard of care in the NHS from baseline across all available timepoints | From baseline up to 60 months
Pharmacokinetic (PK) parameter: Cmax of IPN60130 | From baseline up to Month 24
  Cmax is defined as the maximum observed concentration of IPN60130
PK parameter: AUC of IPN60130 | Every 6 months up to Month 24
  AUC is defined as the concentration of drug over time.
PK parameter: Ctrough of IPN60130 | Every 6 months up to Month 24
  Ctrough is defined as the plasma concentration at the end of the dosing interval.
PK parameter: Cmin of IPN60130 | Every 6 months up to Month 24
  Cmin is defined as the minimum observed concentration of IPN60130
Assessment of the exposure-response relationship | From baseline up to 60 months
  The exposure-response relationship will be assessed by modelling using relevant efficacy and safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (25):
- United States (4):
  - University of California San Francisco (UCSF), San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Perelman School of Medicine - The University of Pennsylvania, Philadelphia, Pennsylvania
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Royal North Shore Hospital - New South Wales, Sydney, Australia
- University Hospitals Leuven, Leuven, Belgium
- Canada (2):
  - University of Alberta, Alberta Health Services (AHS), Edmonton
  - University Health Network (UHN), Toronto General Hospital (TGH), Toronto
- China (4):
  - Children's Hospital Capital Institute of Pediatrics (CIP), Beijing
  - Peking Union Medical College Hospital, Beijing
  - Shangai Children Medical Center, Shanghai
  - Tongi University - Tongi Hospital, Shanghai
- France (2):
  - Groupe Hospitalier Necker Enfants Malades, Paris
  - Hopital Lariboisiere, Paris
- Irccs Gaslini Institute, Genoa, Italy
- Japan (3):
  - Nagoya University Hospital, Nagoya
  - Aichi Children's Health and Medical Center, Ōbu
  - The University of Tokyo Hospital, Tokyo
- Instituto Nacional De Rehabilitacion, Mexico City, Mexico
- Hospital Center Lisbon North, E.P.E- Hospital Santa Maria, Lisbon, Portugal
- Seoul National University Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Universitario Ramon y Cajal, Pozuelo de Alarcón
  - Hospital Universitario Y Politecnico La Femerge, Valencia
- Norrlands Universitetssjukhus, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/